CLINICAL TRIAL: NCT07174778
Title: The Effects of Episodic Future Thinking in Promoting Adherence to Anticoagulation Among Patients With Atrial Fibrillation: a Randomized Controlled Trail
Brief Title: Episodic Future Thinking to Improve Anticoagulant Adherence in Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiawen You (Other)
Responsible Party: Sponsor-Investigator, Jiawen You, Postgraduate student, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L2025SYSU-HL-022
Record Dates: First submitted 2025-09-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Stroke; Episodic Future Thinking; Delay Discounting
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic future thinking (Experimental): Participants will generate individualized episodic future events and transform them to text-based and picture-based cues which will reminder participants to re-imagine their future events in their daily life.
  Interventions: Behavioral: Episodic future thinking
- Attention control (Placebo Comparator): Researchers will maintain equal contact frequency with controls, limited to general check-in messages.
  Interventions: Behavioral: attention control

INTERVENTIONS:
Behavioral: Episodic future thinking — Participants will engage in episodic future thinking prompted via text-based cues and picture-based cues to help them adhere to oral anticoagulants. Participants will also receive health education on atrial fibrillation-related stroke prevention.
  Arms: Episodic future thinking
Behavioral: attention control — The control group will receive standard care, including routine health education from ward nurses and one post-discharge telephone follow-up. In additon, participants will receive a message from the researcher at the same time point each day, but the message will only involve daily greetings.
  Arms: Attention control

SUMMARY:
The purpose of this study is to assess the effectiveness of Episodic Future Thinking (EFT) on improving medication adherence in atrial fibrillation (AF) patients taking oral anticoagulants. A total of 68 participants will be randomly assigned to the intervention group or the control group. Those in the intervention group will receive a 3-week EFT intervention in addition to the usual care, while those in the control group will receive the usual care only. Data on medication adherence, delay discounting (DD), and anticoagulation knowledge will be collected at baseline, end of intervention, and 3-month follow-up.

DETAILED DESCRIPTION:
Participants (N = 68) will be randomly assigned to either an episodic future thinking (EFT) group or attention control group. We will use stratified block randomization. The randomization will be stratified by study site. Within each site, participants will be randomly assigned to either the intervention or control group in a 1:1 ratio using a computer-generated random allocation sequence with variable block sizes (e.g., 4 and 6). A research assistant not involved in recruitment or assessment will generate the sequence. To ensure allocation concealment, sequentially numbered, opaque, sealed envelopes will be prepared according to the generated sequence. After obtaining consent and confirming eligibility, the enrolling investigator will open the next consecutive envelope in the presence of the participant to assign them to a group.

Participants in the intervention group will receive episodic future thinking intervention in addition to the routine health care. The intervention consists of three sessions. In session 1 (on discharge day), the researcher will first provide face-to-face health education on atrial fibrillation-related stroke prevention and a video on the same topics for participants. The health education cover four topics: 1) definition and causes of atrial fibrillation; 2) atrial fibrillation and stroke risk; 3) anticoagulation therapy for stroke prevention; 4) management of comorbidities and risk factors of atrial fibrillation.Then, participants will be instructed to generate individualized episodic future events by visualizing events that will happen or be planned to happen in the coming 1, 3, 6, and 12 months respectively. Participants will be guided to think the long-term impacts (including the benefits and consequences) of adhering or not adhering to oral anticoagulants on their health when imagining future scenario events. The detailed future scenario events imagined by the participants will be condensed into brief narrative statements and also matched with pictures to form text-based and picture-based cues respectively. During Session 2 (weeks 1-3 post-discharge), researchers will administer these cues to participants via WeChat, with two cues per day for the first week followed by one cue per day for the week 2 to week 3. Participants will be asked to complete episodic future thinking task by re-imagining the episodic event based on the content of the cues received within 24 hours. A total of three reminders including a first message reminder within six hours and a second message within 12 hours will be sent to participants to remind them complete the task if no response received in the required time frame. A nonresponse will be recorded if participants did not complete the task 24 hours later the first prompt was sent. Participants will be also encouraged to practice EFT to enhance their adherence to anticolagulation by themselves at home. Participants in the intervention group also will receive weekly education on atrial fibrillation-related stroke prevention. The topics of education are the same with the first session, with topic 1-2 for week 1, topic 3 for week 2, and topic 4 for week 3. In session 3 ( follow-up after the intervention), participants will be followed up once a month by researchers via WeChat or telephone. During each follow-up, adherence to oral anticoagulant will be assessed and issues relating to the management of the illness will be identified and addressed. Any emergent conditions such as major bleeding relating to anticoagulation will be referred to physicians.

The control group will receive usual care, including brief information on atrial fibrilation from ward nurses and one post-discharge telephone follow-up. To reduce potential attention bias, the control group will receive greeting calls from researcher during follow-up with same frequency as the intervention group. In each greeting call, the research will only make greetings or give general information on the illness to participants, no health education will be delivered, and health problems will be addressed.

Data on adherence to anticoagulation, delay discounting and anticoagulation knowledge will be collected at baseline (T0), immediately after the intervention (T1), as well at 3-month follow up (T2). Trained outcome assessors, blinded to group allocation and independent of all other trial procedures, will perform all endpoint evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for atrial fibrillation per the Chinese Guidelines for the Diagnosis and Management of Atrial Fibrillation, with clinically stable condition
* Current or previous use of oral anticoagulants
* Age ≥18 years
* Capable of using WeChat mobile application
* Willing to provide informed consent

Exclusion Criteria:

* Comorbid severe impairment of major organ systems or end-stage disease
* Significant visual or auditory impairments
* Documented cognitive dysfunction or psychiatric disorders (e.g., major depressive disorder, schizophrenia, bipolar disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | Baseline, 3 weeks and 15 weeks
  This study assessed oral anticoagulant adherence using the General Medication Adherence Scale (GMAS) . The 11-item scale evaluates three dimensions: (1) patient behavior related non-adherence (five items), (2) additional disease and pill burden (four items) and (3) cost-related non-adherence (two items). Each item is rated on the scale that 0 = always, 1 = mostly, 2 = sometimes, and 3 = never. Higher scores indicate better adherence and it was divided into five levels according to different scores: 30-33 (high adherence), 27-29 (good adherence), 17-26 (moderate adherence), 11-16 (low adherence), and 0-10 (poor adherence).

SECONDARY OUTCOMES:
Delay discounting for money | Baseline, 3 weeks, 15 weeks
  Delay discounting for money was measured through the Monetary Choice Questionnaire (MCQ). In this test, participants were asked to make a series of choices between smaller-immediate and larger-delayed hypothetical monetary rewards. An example of a question is "Would you prefer $54 today, or $55 in 117 days?". Based on the participants' responses, the delay discounting rate (k) can be calculated. Higher k values indicate a pattern for choosing the rewards in the proximal time frame. All monetary options presented in the questionnaire are entirely hypothetical scenarios. They are designed solely to measure participants' decision-making preferences in an imagined context and do not, in any way, represent the actual compensation or rewards that will be paid to participants in this study.
Delay discounting for health | Baseline, 3 weeks and 15 weeks
  A self-developed Health Intertemporal Choice Questionnaire was used to measure individual delay discounting rates for health outcomes. Patients with atrial fibrillation were presented with a series of choices between a near-term option-"X% reduction in stroke risk after one month of oral anticoagulant therapy"-and a delayed option-"a 65% reduction in stroke risk after one year of oral anticoagulant therapy." The value of Y in the delayed option was fixed at 65%, while the near-term option X ranged from 5% to 60%, increasing in increments of 5%. An example of a question is "Which would you prefer: a 5% reduction in stroke risk after one month of oral anticoagulant use, or a 65% reduction in stroke risk after one year of oral anticoagulant use?"
Anticoagulation knowledge | Baseline, 3 weeks, 15 weeks
  The Anticoagulation Knowledge Tool (AKT) was employed to measure participants' anticoagulation knowledge. The AKT assesses five domains: basic drug information, adverse effects, therapeutic monitoring, drug interactions, and dietary considerations. Section I (20 items) evaluates knowledge of both novel oral anticoagulants and warfarin, while Section II (8 items) focuses specifically on warfarin. Only Section I was utilized in this study.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Gangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Gangdong

IPD SHARING:
Plan to Share IPD: No